CLINICAL TRIAL: NCT04032587
Title: Modification of Pavlovian and Instrumental Learning in Human Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anne Beck, Dr. rer. medic. Dipl.-Psych., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRR265 C02
Record Dates: First submitted 2019-07-18; First posted 2019-07-25 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Alcohol Use Disorder (Mild vs. Moderate to Heavy)
Keywords: approach / avoidance; alcohol use disorder; stress; stress reduction; goal-directed decision-making
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-treatment seeking subjects with Alcohol Use Disorder (Experimental): AUD; mild vs. moderate to heavy
  Interventions: Behavioral: Modified training version of the Approach / Avoidance Task (AAT, see Wiers et al., 2011); Behavioral: Mindfulness-based interventions (e.g. body scan)
- Healthy Controls (Active Comparator)
  Interventions: Behavioral: Modified training version of the Approach / Avoidance Task (AAT, see Wiers et al., 2011); Behavioral: Mindfulness-based interventions (e.g. body scan)

INTERVENTIONS:
Behavioral: Modified training version of the Approach / Avoidance Task (AAT, see Wiers et al., 2011) — First, a modified training version of the Approach Avoidance Task, (see Wiers et al. 2011) with arbitrary Pavlovian cues will be developed and the effectiveness of this manipulation will be assessed. In detail, positive as well as negative Pavlovian cues (derived from a Pavlovian-to-Instrumental transfer Task, see Garbusow et al. 2014, Garbusow et al. 2016) will be modified according to their approach/ avoidance propensities by 1) approaching negative stimuli (pulling joystick), 2) approaching positive stimuli (pulling joystick), 3) avoiding negative stimuli (pushing joystick) and 4) avoiding positive stimuli (pushing joystick). Thus, we aim at reversing the PIT effect (pushing positive cues/ pulling negative cues) or enhancing the PIT effect (pulling positive cues/ pushing negative cues).
Behavioral: Mindfulness-based interventions (e.g. body scan) — Acute stress reduction will be applied in a standardized way using audio files with an anticipated duration of 20-30 minutes.

SUMMARY:
The project aims at investigating modifications of environmental factors (i.e. cues and stress) relevant for learning mechanisms in addictive disorders.

DETAILED DESCRIPTION:
Project C02 aims at investigating modifications of environmental factors (i.e. cues and stress) relevant for learning mechanisms in addictive disorders. The investigators will examine non-treatment seeking subjects with alcohol use disorder (AUD; mild vs. moderate to heavy), and healthy controls with a focus on the impact of Pavlovian conditioned stimuli (context-related cues) on instrumental behavior (so-called Pavlovian-to-Instrumental transfer (PIT)) and whether the PIT effect can be systematically modified by manipulating the approach/ avoidance propensities of Pavlovian cues (work package (WP) 1). Concerning stress as a major modulator of cue reactivity in addiction, the investigators further plan to assess whether acute, active stress reduction modifies such PIT effects (i.e. decreasing transfer effects) as well as goal-directed vs. habitual behavior (i.e. strengthening goal-directed decisionmaking) (WP2). Lastly, this project aims at contributing to the understanding of the underlying neurobiological correlates of manipulation of approach/ avoidance propensities of Pavlovian cues and acute stress reduction by using functional magnetic resonance imaging (WP3) with a focus on amygdala-striatal activity (PIT) and frontostriatal processes (goaldirected decision-making).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 16-32 years, 33-49 years, and aged 50-65 years
2. Mild, moderate to heavy alcohol-use disorder (AUD) according to DSM-5 criteria (mild: 2-3 AUD criteria; moderate: 4-5 AUD criteria; heavy: 6 or more AUD criteria); not clinically requiring detoxification (as confirmed by an independent board-certified psychiatrist); AUD patients can have mild to moderate cannabis use disorder as well as tobacco use disorder
3. Ability to provide fully informed consent and to use self-rating scales
4. Willingness to use an android phone
5. Sufficient understanding of the German language

Exclusion Criteria:

1. Lifetime history of DSM-5 bipolar disorder, schizophrenia or schizophrenia spectrum disorder, or substance dependence other than alcohol or nicotine or cannabis dependence. Severe alcohol and cannabis use disorder will be excluded.
2. Current threshold DSM-5 diagnosis of major depressive disorder, or presence of suicidal intention
3. History of severe head trauma or other severe central nervous system disorder (e.g., dementia, Parkinson's disease, multiple sclerosis)
4. Pregnancy or nursing infants
5. Current use of medications or drugs known to interact with the CNS within at least four half-life post last intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent especially within the ventral striatum and the amygdala (fMRI) | 2 consecutive days
Rate of Pavlovian-to-instrumental-Transfer (instrumental responding, i.e.number of button presses, in dependence of Pavlovian Stimuli) | 2 consecutive days
Rate of goal-directed decision-making/habitual decision making | 2 consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Psychiatry, CCM, Charite Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Beck A, Schlagenhauf F, Wustenberg T, Hein J, Kienast T, Kahnt T, Schmack K, Hagele C, Knutson B, Heinz A, Wrase J. Ventral striatal activation during reward anticipation correlates with impulsivity in alcoholics. Biol Psychiatry. 2009 Oct 15;66(8):734-42. doi: 10.1016/j.biopsych.2009.04.035. Epub 2009 Jun 27. PMID 19560123
- [Background] Beck A, Wustenberg T, Genauck A, Wrase J, Schlagenhauf F, Smolka MN, Mann K, Heinz A. Effect of brain structure, brain function, and brain connectivity on relapse in alcohol-dependent patients. Arch Gen Psychiatry. 2012 Aug;69(8):842-52. doi: 10.1001/archgenpsychiatry.2011.2026. PMID 22868938
- [Background] Beck A, Pelz P, Lorenz RC, Charlet K, Geisel O, Heinz A, Wustenberg T, Muller CA. Effects of high-dose baclofen on cue reactivity in alcohol dependence: A randomized, placebo-controlled pharmaco-fMRI study. Eur Neuropsychopharmacol. 2018 Nov;28(11):1206-1216. doi: 10.1016/j.euroneuro.2018.08.507. Epub 2018 Sep 11. PMID 30217552
- [Background] Beylergil SB, Beck A, Deserno L, Lorenz RC, Rapp MA, Schlagenhauf F, Heinz A, Obermayer K. Dorsolateral prefrontal cortex contributes to the impaired behavioral adaptation in alcohol dependence. Neuroimage Clin. 2017 Apr 17;15:80-94. doi: 10.1016/j.nicl.2017.04.010. eCollection 2017. PMID 28491495
- [Background] Friedel E, Schlagenhauf F, Beck A, Dolan RJ, Huys QJ, Rapp MA, Heinz A. The effects of life stress and neural learning signals on fluid intelligence. Eur Arch Psychiatry Clin Neurosci. 2015 Feb;265(1):35-43. doi: 10.1007/s00406-014-0519-3. Epub 2014 Aug 21. PMID 25142177
- [Background] Genauck A, Quester S, Wustenberg T, Morsen C, Heinz A, Romanczuk-Seiferth N. Reduced loss aversion in pathological gambling and alcohol dependence is associated with differential alterations in amygdala and prefrontal functioning. Sci Rep. 2017 Nov 24;7(1):16306. doi: 10.1038/s41598-017-16433-y. PMID 29176580
- [Background] Koehler S, Ovadia-Caro S, van der Meer E, Villringer A, Heinz A, Romanczuk-Seiferth N, Margulies DS. Increased functional connectivity between prefrontal cortex and reward system in pathological gambling. PLoS One. 2013 Dec 19;8(12):e84565. doi: 10.1371/journal.pone.0084565. eCollection 2013. PMID 24367675
- [Background] Koehler S, Hasselmann E, Wustenberg T, Heinz A, Romanczuk-Seiferth N. Higher volume of ventral striatum and right prefrontal cortex in pathological gambling. Brain Struct Funct. 2015 Jan;220(1):469-77. doi: 10.1007/s00429-013-0668-6. Epub 2013 Nov 16. PMID 24240601
- [Background] Romanczuk-Seiferth N, Koehler S, Dreesen C, Wustenberg T, Heinz A. Pathological gambling and alcohol dependence: neural disturbances in reward and loss avoidance processing. Addict Biol. 2015 May;20(3):557-69. doi: 10.1111/adb.12144. Epub 2014 Apr 22. PMID 24754423
- [Background] Seo S, Mohr J, Beck A, Wustenberg T, Heinz A, Obermayer K. Predicting the future relapse of alcohol-dependent patients from structural and functional brain images. Addict Biol. 2015 Nov;20(6):1042-55. doi: 10.1111/adb.12302. Epub 2015 Oct 4. PMID 26435383